CLINICAL TRIAL: NCT02747550
Title: Temporary Simultaneous Two-arterial Occlusions to Reduce Operative Blood Loss During Laparoscopic Myomectomy: a Randomized Controlled Trial
Brief Title: Temporary Simultaneous Two-arterial Occlusions During Laparoscopic Myomectomy
Acronym: TESTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-04-053
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Myoma
MeSH Terms: conditions — Myoma | interventions — testo

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LM with TESTO (Experimental): In subjects allocated to the experimental group, the temporary simultaneous two-arterial occlusions (TESTO) procedure was performed to minimize operative blood loss during laparoscopic myomectomy.
  Interventions: Procedure: LM with TESTO
- LM without TESTO (Active Comparator): In the control group, no intervention for the temporary simultaneous two-arterial occlusions (TESTO) procedure was made during laparoscopic myomectomy.
  Interventions: Procedure: LM without TESTO

INTERVENTIONS:
Procedure: LM with TESTO — In subjects allocated to the experimental group, the temporary simultaneous two-arterial occlusions (TESTO) procedure was performed to minimize operative blood loss during laparoscopic myomectomy.
  Arms: LM with TESTO
Procedure: LM without TESTO — In the control group, no intervention for the temporary simultaneous two-arterial occlusions (TESTO) procedure was made during laparoscopic myomectomy
  Arms: LM without TESTO

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of the temporary simultaneous two-arterial occlusions (TESTO) on operative blood loss during laparoscopic myomectomy.

DETAILED DESCRIPTION:
Significant hemorrhage is major perioperative concern in myomectomy, and can result in need of blood transfusion, conversion to hysterectomy, development of hypovolemic shock and postoperative anemia, and delayed recovery. Therefore, methods to decrease operative blood loss during myomectomy in women wishing to preserve their uterus and fertility are important and must be developed.

ELIGIBILITY:
Inclusion Criteria:

* women with symptomatic myomas such as menorrhagia, pelvic pressure/pain, or infertility
* women who were planning to undergo laparoscopic myomectomy
* women who had ≤ 10 myomas, with the largest myoma ≤ 10 cm
* women with regular menstrual bleeding
* women who were not pregnant at the surgery
* women between 19 and 48 years of age.

Exclusion Criteria:

* women who underwent concomitant complex surgical procedures at the time of laparoscopic myomectomy, such as severe adhesiolysis or resection for severe endometriosis
* women who were in postmenopausal or climacteric status
* women with a history of oophorectomy or salpingo-oophorectomy
* women with any suggestion of malignant uterine or adnexal diseases
* women with major medical comorbidities or psychiatric illnesses, which could affect follow-up and/or compliance
* women who refused to participate or give consent to the procedures

Ages: 19 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
operative blood loss | the day of surgery
  Operative blood loss was calculated by the anesthesiology unit as the difference between the total amount of suction and irrigation plus the difference between the total gauze weight before and after surgery.

SECONDARY OUTCOMES:
change in hemoglobin | post-operative day 1
  The change in hemoglobin change was defined as the difference between the preoperative hemoglobin level and the hemoglobin level on postoperative day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD, PhD, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No